CLINICAL TRIAL: NCT07164820
Title: The Effect of Su Jok Therapy on Pain During Heel LanceProcedure in Newborn
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ayse Aydin, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Büşra KORKMAZ
Record Dates: First submitted 2025-08-31; First posted 2025-09-10 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Heel Lance Procedures; Pain Management
Keywords: pain; heel lance procedures; Su Jok Therapy; newborn
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Statistics expert, Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Su Jok Therapy (Experimental): For newborns who meet the inclusion criteria, the Data Collection Form and the Neonatal Pain, Agitation, and Sedation Scale (N-PASS) will be completed prior to the procedure.
  Following the completion of these forms, Su Jok therapy will be applied for 5 minutes.
  Subsequently, a heel lance procedure will be performed. During and after the procedure, pain assessment will be conducted using the N-PASS.
  Interventions: Other: Su Jok Application
- Routine Heel Lance (No Intervention): For newborns who meet the inclusion criteria, the Data Collection Form and the Neonatal Pain, Agitation, and Sedation Scale (N-PASS) will be completed prior to the procedure.
  Following the completion of these forms, routine heel lance will be performed. During and after the procedure, pain assessment will be conducted using the N-PASS.

INTERVENTIONS:
Other: Su Jok Application — Description: The newborn's hands will be used for the application. Su Jok therapy will be administered by applying massage and seeds to the corresponding reflection points on the hand prior to the he
  Arms: Su Jok Therapy

SUMMARY:
Objective: To determine the effect of Su Jok therapy on pain levels during the heel lance procedure in newborns. The study will be conducted as a randomized controlled experimental trial with a pretest-posttest control group design. The heel lance procedure will be video recorded, and pain assessment will be performed independently by an experienced neonatal intensive care nurse with 7 years of clinical expertise and a neonatologist, using validated pain assessment scales.

DETAILED DESCRIPTION:
This study aims to examine the effect of Su Jok therapy on pain experienced during the heel lance procedure in newborns. Reducing pain associated with heel lance, one of the most commonly performed invasive procedures in the neonatal period, is crucial for the health and comfort of infants. Su Jok therapy is a non-invasive and side-effect-free method applied by stimulating specific points on the hands and feet, and in this study, it is considered as an alternative approach for pain management during heel lance procedures.

The research will be conducted between July 1, 2025, and July 1, 2026, in Family Health Centers affiliated with the Rize Provincial Health Directorate. A total of 66 term newborns (≥37 gestational weeks), consisting of 33 infants in the intervention group and 33 infants in the control group, will be included. The study sample size was determined using G\*Power 3.1.9.7 software. Based on a two-group (experimental, control) and three-measurement (pretest, procedure test, posttest) design with Two-Way Mixed ANOVA analysis, an effect size of 0.20 (f = 0.20), an alpha of 0.05, and a power of 90% (1-β = 0.90) were used, resulting in a required sample of 28 per group. Considering potential data loss, the sample size was increased by 20% per group, leading to a final sample size of 33 per group, 66 in total.

**Inclusion criteria:**

* Term newborns (≥37 gestational weeks)
* Without neurological disorders
* Who have not undergone any painful procedure (e.g., injection, venipuncture) in the previous 24 hours
* For whom heel lance for routine screening tests is planned
* Whose parents provided written informed consent
* Who have not received analgesic or sedative medications

**Exclusion criteria:**

* Clinically unstable infants before or during the procedure (e.g., respiratory distress, cardiac instability)
* Infants whose position was changed, intervention was interrupted, or procedure repeated in a way that could affect pain perception
* Parental withdrawal of consent during the procedure
* Severe restlessness or sudden physiological changes preventing pain assessment
* Infants for whom standardized data could not be collected due to protocol violations

From eligible newborns presenting to the centers during the study period, 66 infants will be randomly selected according to the sample size determined by power analysis. Using randomization software, 33 newborns will be assigned to the intervention group and 33 to the control group. Randomization will minimize bias in group allocation. Due to the nature of the study, blinding of the researcher will not be possible; however, blinding will be applied to participants and the statistician. Parents will not know the group allocation of their infants. After the study is completed, coded data from both groups (Group A and Group B) will be analyzed by an independent statistician to ensure objectivity. Thus, the study is planned as a double-blind randomized controlled trial.

**Data collection tools:**

1. **Newborn Introductory Information Form** - prepared by the researcher, including demographic and clinical data (Apgar score, gender, weight, height, head circumference, feeding method). It also records heart rate, oxygen saturation, and crying duration before, during, and after the procedure.
2. **Neonatal Pain/Agitation and Sedation Scale (N-PASS)** - developed for use in all neonates, both term and preterm. It can be used to assess both acute and chronic pain, as well as in infants receiving mechanical ventilator support. The scale includes five subdimensions: crying/irritability, behavior, facial expression, extremity tone, and vital signs. In this study, only the pain/agitation section will be used.

**Intervention procedure:** Newborns meeting inclusion criteria will first undergo baseline data collection (Introductory Information Form and N-PASS). In the intervention group, Su Jok therapy will be applied for 5 minutes immediately before heel lance. The procedure consists of gentle circular massage with mild pressure on specific reflex points on the hand by the researcher, while the newborn is kept in a comfortable position. After the intervention, heel lance will be performed, and pain will be assessed during and after the procedure using N-PASS.

In the control group, baseline forms will be completed, and routine heel lance will be performed without any Su Jok intervention. Pain will be assessed during and after the procedure with N-PASS.

Environmental conditions (room temperature 32-34°C, minimal lighting and noise) will be standardized. Sterile and hygienic practices will be followed, with strict hand hygiene before each application. In both groups, pain assessments will be supported by monitoring heart rate, oxygen saturation, and recovery time. All procedures will prioritize neonatal comfort, safety, and ethical compliance.

ELIGIBILITY:
Inclusion Criteria:

* Term newborns (≥37 gestational weeks)
* Without neurological disorders
* Who have not undergone any painful procedure (e.g., injection, venipuncture) in the previous 24 hours
* For whom heel lance for routine screening tests is planned
* Whose parents provided written informed consent
* Who have not received analgesic or sedative medications

Exclusion Criteria:

* Clinically unstable infants before or during the procedure (e.g., respiratory distress, cardiac instability)
* Infants whose position was changed, intervention was interrupted, or procedure repeated in a way that could affect pain perception
* Parental withdrawal of consent during the procedure
* Severe restlessness or sudden physiological changes preventing pain assessment
* Infants for whom standardized data could not be collected due to protocol violations

Ages: 1 Day to 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Neonatal Pain/Agitation and Sedation Scale (N-PASS) | 12 months
  The Neonatal Pain/Agitation and Sedation Scale (N-PASS) was developed by Hummel et al. in 2003 for use in all neonates, both term and preterm. A further advantage of the N-PASS is that it can be used to assess both acute and chronic pain, as well as in infants receiving mechanical ventilator support. The scale was revised by Pat Hummel on October 2, 2009 (Hummel et al., 2008; Hummel et al., 2010). The Turkish adaptation of the scale was performed by Açıkgöz et al. in 2011, who reported Cronbach's Alpha internal consistency coefficients of 0.797 for the pre-procedure period and 0.917 for during and post-procedure.
  The scale consists of two distinct sections: one for assessing the level of sedation and another for the level of pain. The N-PASS comprises five sub-parameters. These are: crying and irritability, behavior/state, facial expression, extremities (arms/legs) and trunk tone, and vital signs. In pain assessment, each behavioral and physiological criterion
Neonatal Introductory Information Form | 12 months
  This form was developed by the researcher and includes introductory questions regarding the newborn.
  The Neonatal Introductory Information Form contains items such as Apgar score, sex, weight, length, head circumference, feeding type, and feeding route.
  In addition, it includes a section designed to record the newborn's heart rate, oxygen saturation, and crying duration before, during, and after the heel lance procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe AYDIN, Study Director — Ataturk University
Locations (1):
- ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No